CLINICAL TRIAL: NCT01436539
Title: A Multi-center, Open Label, Randomized Study of Effects and Safety Between Adefovir Dipivoxil Plus Polyene Phosphatidylcholine Capsule Versus Adefovir Dipivoxil Alone in Chronic Hepatitis B Patients
Brief Title: Study of Effects and Safety Between Adefovir Dipivoxil Plus Polyene Phosphatidylcholine Versus Adefovir Dipivoxil Alone in Chronic Hepatitis B Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jun Cheng (Other)
Collaborators: Sanofi (Industry); Fujian Cosunter Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor-Investigator, Jun Cheng, Vice president, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ditan-2011-01
Record Dates: First submitted 2011-09-13; First posted 2011-09-19 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir dipivoxil; polyene phosphatidylcholine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adefovir Dipivoxil and polyene phosphatidylcholine (Experimental): Adefovir Dipivoxil 10 mg once daily for 48 weeks plus Polyene phosphatidylcholine (PPC) 456 mg three times per day for 48 weeks
  Interventions: Drug: Adefovir Dipivoxil and polyene phosphatidylcholine
- Adefovire Dipivoxil (Active Comparator): Adefovir Dipivoxil 10 mg once daily for 48 weeks
  Interventions: Drug: Adefovir Dipivoxil

INTERVENTIONS:
Drug: Adefovir Dipivoxil and polyene phosphatidylcholine — Adefovir Dipivoxil 10 mg once daily for 48 weeks plus Polyene phosphatidylcholine (PPC) 456 mg three times per day for 48 weeks
  Arms: Adefovir Dipivoxil and polyene phosphatidylcholine
Drug: Adefovir Dipivoxil — Adefovir Dipivoxil 10 mg once daily for 48 weeks
  Arms: Adefovire Dipivoxil

SUMMARY:
The purpose of the study is to evaluate the effects and safety of Adefovir Dipivoxil plus polyene phosphatidylcholine compared to Adefovir Dipivoxil alone in patients with chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the age of 18 to 65 years with chronic hepatitis B.
* HBsAg positive for a minimum of 6 months.
* HBV DNA ≥4 log10 copies/ml, and ≤ 6 log10 copies/mL
* Alanine aminotransferase (ALT) ≥ 2 times the upper limit of normal(ULN) and ≤10 times ULN, and documented ALT abnormal within 6 month prior to the study screening.
* Had a liver biopsy performed within 6 months prior to randomization and has readable biopsy slides or agrees to have a biopsy performed prior to entry.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Received any nucleoside, nucleotide or interferon therapy within 6 months prior to the screening.
* Previous treatment with lamivudine, adefovir, entecavir or telbivudine and occurred viral breakthrough or genotype resistance.
* Received immunosuppressive agents or other immunoregulates (including thymosin),systemic cytotoxic drugs, other antiviral agents including Chinese herb medicine within 6 months prior to the screening.
* Active alcohol intake( more than 20g/d for female or more than 30g/d for male) or drug abuse within 1 year prior to screening. Alcohol or drug abuse considered by the investigator to be sufficient to hinder compliance with treatment, participation in the study or interpretation of results.
* ALT is greater than 10 times ULN at screening or has the history of transient decompensated liver disease due to acute exacerbation.
* Any of the laboratory test at screening as the following :

  * serum creatinine > 1.5 mg/dl ;
  * prothrombin time ≥ 4 seconds prolonged or PTA <60%;
  * serum albumin<32 g/L;
  * serum bilirubin>3.0mg/dL;
  * Hemoglobin<11g/dL(males) or <10 g/dL(females), white blood cells count<3.5 x 10^9/L, absolute neutrophil count <1.5 x 10^9/L, platelets<80 x 10^9/L.
* Patient is coinfected with HCV, HDV or HIV.
* Hepatocellular carcinoma (HCC), or the presence of a mass on imaging studies of the liver that is suggest of HCC, or an alpha-fetoprotein (AFP)> 500ng/mL.
* Decompensated liver disease as defined by serum bilirubin >3mg/dL, prothrombin time≥ 4 seconds prolonged, a serum albumin<32g/L, or a history of ascites, variceal bleeding or hepatic encephalopathy.
* Presence of other causes of liver disease (i.e.alcoholic liver disease,autoimmune hepatitis, hemochromatosis, Wilson disease, nonalcoholic steatohepatitis, alpha-1anti-trypsin deficiency).
* Any serious or active medical or psychiatric illnesses other than hepatitis B which, in the opinion of the investigator, would interfere with patient treatment, assessment or compliance with the protocol. This would include, may not limit to, renal, cardiac, pulmonary, vascular, neurogenic, digestive, metabolic (diabetes, thyroid disorders, adrenal disease), immunodeficiency disorders, active infection or cancer.
* BMI≥30.
* Patient is pregnant or breast-feeding.
* Planned for liver transplantation or previous liver transplantation.
* Need take hepatotoxic drugs (e.g.,dapsone, erythromycin, fluconazole, rifampin, etc) and nephrotoxic drugs (e.g., NSAIDs, aminoglycosides, amphotericin B, foscarnet, etc.) for long time.
* History of hypersensitivity to nucleoside analogues.
* Previous (or planned) participation in an investigational trial involving administration of investigational compound within 12 weeks prior to the study screening.
* Poor compliance of the patient considered by investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-03 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Proportions of subjects with histological response in treatment and control group. | at week 48

SECONDARY OUTCOMES:
Proportions of subjects in each group who achieve: HBV DNA < 300 copies/mL | at week 48
Mean log10 reduction from baseline in HBVDNA | at week 12, 24, 48
ALT normalization rate and range | at week 12 and 48
Liver stiffness values reduction from baseline by Fibroscan | at week 48
HBeAg loss and HBe seroconversion | at week 12 and 48
HBsAg loss and HBs seroconversion | at week 12 and 48
Improvement in symptoms score | at week 12, 24 and 48
Frequency of adverse events | up to 60 weeks
Frequency of serious adverse events | up to 60 weeks
Frequency of discontinuations from study drug due to adverse events or laboratory abnormalities. | up to 60 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan Hospital, Capital Medical University, Beijing, China